CLINICAL TRIAL: NCT07278544
Title: Harnessing Communication Preferences to Enhance Its Persistence and Mitigate Relapse of Challenging Behavior
Brief Title: Harnessing Communication Preferences
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joel E. Ringdahl (Other)
Collaborators: University of Iowa (Other); University of Florida (Other); Virginia Polytechnic Institute and State University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Joel E. Ringdahl, Professor, University of Georgia
Organization: University of Georgia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VERSION00004073; 2R01HD069377-12A1 (NIH)
Record Dates: First submitted 2025-08-27; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Intellectual Disability; Autism Spectrum Disorder; Self-Injurious Behavior; Communication Disabilities; Communication, Nonverbal
Keywords: Functional communication training; Treatment maintenance; Behavioral relapse
MeSH Terms: conditions — Intellectual Disability; Autism Spectrum Disorder; Self-Injurious Behavior; Communication Disorders; Nonverbal Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrefFCT (Experimental): PrefFCT involves reinforcing an appropriate communicative response determined to be preferred by the individual relative to a second appropriate communicative response. During PrefFCT, participants will receive access to the functionally relevant reinforcer following occurrences of the specified communication modality. Challenging behavior will not produce any programmed consequence.
  Interventions: Behavioral: PrefFCT
- NonPrefFCT (Experimental): NonPrefFCT involves reinforcing an appropriate communicative response determined to be less preferred by the individual relative to another appropriate communicative response. During NonPrefFCT, participants will receive access to the functionally relevant reinforcer following occurrences of the specified communication modality. Challenging behavior will not produce any programmed consequence.
  Interventions: Behavioral: NonPrefFCT

INTERVENTIONS:
Behavioral: PrefFCT — Differential reinforcement of alternative communication and extinction of challenging behavior.
  Arms: PrefFCT
Behavioral: NonPrefFCT — Differential reinforcement of alternative communication and extinction of challenging behavior.
  Arms: NonPrefFCT

SUMMARY:
The goal of this clinical trial is to evaluate how preference for communication approach (e.g., using a touch talker versus picture cards) impacts treatment maintenance in the context of treatment to reduce challenging behavior exhibited by individuals with intellectual and/or developmental disabilities. As well, the clinical trial will evaluate how this preference impacts treatment relapse when care providers implement intervention and will identify potential demographic variables (e.g., age and symptom severity) that affect outcomes.

The main question[s] it aims to answer [is/are]:

Preferred communication strategies will persist to a greater extent when intervention is disrupted, relative to less preferred communication strategies.

Communication modality preference will increase persistence for individuals with lower pre-experimental symptom severity scores and higher pre-experimental communication functioning scores. We predict demographic characteristics and developmental level will not impact intervention outcomes.

Two groups will be compared. Group 1 will receive initial intervention using a preferred communication strategy. Group 2 will receive initial intervention using a non preferred, but effective, communication strategy. Intervention type will then be reversed. Researchers will compare preferred and non preferred interventions on continued expression of the communication strategy when intervention is challenged.

Participants will exhibit alternative appropriate communicative behavior as a means of replacing/reducing challenging behavior. This will take place using (a) preferred communication strategies and (b) non preferred communication strategies. Following successful intervention with each type of communication, intervention will be challenged and continued use of the communication strategy will be measured.

DETAILED DESCRIPTION:
Participants and Setting

Sixty individuals with IDD who engage in challenging behavior (e.g., aggression, self-injury, property destruction) and have little to no communication will be recruited to participate in this study (we anticipate completion of the project for at least 48 participants). Participants will include those for whom two device-based alternative and augmentative communication (AAC) strategies can be identified.

Pre-Experimental Phase

Prior to randomization, all participants will complete several assessments to establish two different functional-communication modalities that are considered device-based AAC strategies (e.g., picture card, microswitch, tablet app). Initial modalities will be identified through a validated assessment that has been shown to identify proficient communication modalities. Next, the individual's preference will be assessed between those established modalities. These assessments are the same ones conducted in our currently funded study and include a preference assessment among leisure items and activities, a functional analysis of challenging behavior, a communication-modality proficiency assessment, FCT, and a communication-modality preference assessment. From the communication modality preference assessment, a high preferred and lesser preferred modality will be identified. These modalities henceforth will be referred to as follows: preferred communication modality (PrefFCT) and lesser preferred communication modality (NonPrefFCT).

Randomization

Following the completion of all assessments in the pre-experimental phase, participants will be randomized to one of two initial conditions: PrefFCT or NonPrefFCT. Because this is a crossover design, each participant will experience the other modality condition after crossover. Further, participants will also be randomized into their implementer condition (different trained therapist versus trained caregiver) in a similar manner. After random assignment, all participants will undergo the same sequence of procedures but using the communication modality according to condition assignment.

Crossover

Following completion of FCT and disruption after initial randomization, participants will crossover to the alternative condition and complete FCT and disruption with the other communication modality, allowing for within-subjects comparisons. That is, participants who were originally assigned to the PrefFCT condition and completed FCT and disruption with their preferred communication modality will then move to the NonPrefFCT condition during the crossover phase and thus complete a second round of FCT and disruption, but with their lesser preferred communication modality. The opposite will occur for those who started in the NonPrefFCT condition.

ELIGIBILITY:
Inclusion Criteria:

* 2 years old and older.
* Diagnosis of intellectual or developmental disability.
* Referred for assessment and treatment of challenging behavior.

Exclusion Criteria:

* Challenging behavior does not occur within the context of structured assessment, eliminating the ability to identify its operant function, or the behavior is deemed too dangerous to safely observe during assessment.
* Communicate functionally using vocal/verbal communication.
* Can only identify one proficient AAC strategy.

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Persistence of Communication | Change in level of communication from baseline to 6 weeks post baseline.
  Response rate as the average of the communication rate during treatment disruption.

SECONDARY OUTCOMES:
Relapse of Challenging Behavior | Change in level of challenging behavior from baseline to 6 weeks post baseline with new implementer.
  Response rate as the average challenging behavior rate during treatment with new implementer.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Georgia, Athens, Georgia
  - University of Iowa, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: Data will be made available at the time of associated publication or at the end of the performance period, whichever comes first. Data shared in DASH will be preserved for the foreseeable future as DASH does not currently have any data deprecation or sunsetting protocols.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT07278544/ICF_000.pdf